CLINICAL TRIAL: NCT05578729
Title: The Effect of Different Masks Used by Pregnant Women on Vital Signs and Non Stress Test During The COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Yeter ŞENER, Principal Investigator, Bozok University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: YOBU_YETERŞENER_131822
Record Dates: First submitted 2022-10-06; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Covid-19; Pregnant; Fetus; Mask
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Single surgical mask group (n=30) Double surgical mask group (n=30) N95 mask group (n=31)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single surgical mask group (Other): Participants wore single surgical masks.
  Interventions: Behavioral: Single surgical mask group, Double surgical mask group, N95 mask group
- Double surgical mask group (Other): Participants wore double surgical masks.
  Interventions: Behavioral: Single surgical mask group, Double surgical mask group, N95 mask group
- N95 mask group (Other): Participants wore N95 masks.
  Interventions: Behavioral: Single surgical mask group, Double surgical mask group, N95 mask group

INTERVENTIONS:
Behavioral: Single surgical mask group, Double surgical mask group, N95 mask group — Masks were given to the resting pregnant women 30 minutes before the NST, and they were provided to wear masks. After 30 minutes, the vital signs of the pregnant women were measured just before and after the NST, and the images of the NST traces were taken.

SUMMARY:
This study was conducted to examine the effects of different masks used by pregnant women on vital signs and non stress test (NST) during the COVID-19. This study was conducted as a single-blind randomized controlled trial. Healthy pregnant women aged 19 years and older, who were followed up on an outpatient basis, and who were in the 37-40th week of pregnancy, were included in the study. The study consisted of a single surgical mask group (n=30), double surgical mask group (n=30), and N95 mask group (n=31). Masks were given to the resting pregnant women 30 minutes before the NST, and they were provided to wear masks. After 30 minutes, the vital signs of the pregnant women were measured just before and after the NST, and the images of the NST traces were taken.

ELIGIBILITY:
Inclusion Criteria:

1. Being 19 years or older
2. Being pregnant at 37-40 weeks of pregnancy and having healthy pregnancy
3. Being followed on an outpatient basis

Exclusion Criteria:

1. Having a multiple pregnancy
2. Having a systemic, psychiatric disease or psychological problem (thyroid, heart, schizophrenia, etc.)
3. Being in the category of risky pregnancies (Preeclampsia, gestational diabetes, etc.)
4. Smoking
5. Having alcohol and substance use
6. Never done NST before
7. Having an identified risk factor in the fetus
8. Having barriers to communication
9. Being a foreign national
10. Being in contact with, or having, or suspected of having COVID-19 and previously had COVID-19.

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Vital signs | 30 minutes later, just before the NST was performed.
  Blood pressure-Systolic and diastolic (Blood pressure measured in mmHg)
Vital signs | 30 minutes later, just before the NST was performed.
  Respiratory rate (Respiratory rate per minute was measured)
Vital signs | 30 minutes later, just before the NST was performed.
  SpO2 saturation (SpO2 saturation was measured in %)
Vital signs | 30 minutes later, just before the NST was performed.
  Pulse (Pulse was measured in beats per minute/bpm)
Non stress test | Just after the NST was finished (after 20 minutes)
  After the NST was finished, the images were taken by numbering the traces. A folder was created containing the NST traces that were imaged. After all the research data were collected, the NST tracing results (fetal heart rate (bpm), variability, acceleration, deceleration, contraction, reactivity, and non-reactivity) were evaluated by a Gynecology and Obstetrics physician who did not know which group the participants were in.

SECONDARY OUTCOMES:
Vital signs | Just after the NST was finished (after 20 minutes)
  Blood pressure-Systolic and diastolic (Blood pressure measured in mmHg)
Vital signs | Just after the NST was finished (after 20 minutes)
  Respiratory rate (Respiratory rate per minute was measured)
Vital signs | Just after the NST was finished (after 20 minutes)
  SpO2 saturation (SpO2 saturation was measured in %)
Vital signs | Just after the NST was finished (after 20 minutes)
  Pulse (Pulse was measured in beats per minute/bpm)

CONTACTS AND LOCATIONS:
Locations (1):
- Yeter, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I WILL SEND THE JOURNAL AFTER I REGISTER HERE.